CLINICAL TRIAL: NCT05602207
Title: Clinical and Molecular Effects of Abrocitinib in Subjects With Atopic Dermatitis With an Unsatisfactory Response or Facial Erythema After Treatment With Dupilumab
Brief Title: Effects of Abrocitinib in Subjects With Atopic Dermatitis With an Unsatisfactory Response After Treatment With Dupilumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inno-6050
Record Dates: First submitted 2022-07-15; First posted 2022-11-02 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
Keywords: eczema; dupilumab; abrocitinib
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — abrocitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abrocitinib 100 mg tablet (marketed drug) (Experimental)
  Interventions: Drug: Abrocitinib

INTERVENTIONS:
Drug: Abrocitinib — 100 mg Abrocitinib once daily (QD) for 12 weeks
  Other Names: CIBINQO

SUMMARY:
This is a single-arm, open-label study that will examine the effect of abrocitinib in subjects with atopic dermatitis.

DETAILED DESCRIPTION:
This study is being conducted to evaluate the efficacy, safety, and molecular effects of abrocitinib in subjects with an unsatisfactory response or facial erythema after at least 12 weeks of treatment with dupilumab. Approximately 60 subjects with atopic dermatitis will receive abrocitinib once daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject 18 years of age or older, at the time of consent.
2. Subject has clinically confirmed diagnosis of active atopic dermatitis (AD), according to Hanifin and Rajka criteria.
3. Subject has at least a 1-year history of AD and had no significant flares in AD for at least 4 weeks before screening.
4. Subjects who had moderate to severe AD before initiating dupilumab treatment.
5. Subject currently has an unsatisfactory response or facial erythema after at least 12 weeks of treatment with dupilumab, defined as follows:

   1. A global vIGA-AD ≥ 2, at least 1% BSA with facial erythema, and a modified vIGA-AD for the face ≥2 at screening and Day 1 OR
   2. A global vIGA-AD ≥ 2, at least 3% BSA affected by AD on the trunk and/or limbs, and a modified vIGA-AD for the trunk/limbs ≥ 2 at screening and Day 1.

Exclusion Criteria:

1. Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
2. Subject has clinically infected AD.
3. Subject has a history of skin disease or presence of skin condition that would interfere with the study assessments.
4. Subject has a history of cancer within 5 years prior to Day 1.
5. Subject has a history of lymphoproliferative disorder, lymphoma, or leukemia, or signs and symptoms suggestive of current lymphatic or lymphoid disease.
6. Subject has any clinically significant medical condition that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.
7. Subject is known to have immunodeficiency disorder or a first-degree relative with a hereditary immunodeficiency.
8. Subject has a current or recent clinically serious infection.
9. Subject has used abrocitinib prior to Day 1.
10. Subject has a known hypersensitivity to abrocitinib or its excipients.
11. Subject has a known history of clinically significant drug or alcohol abuse within 6 months prior to Day 1 that in the opinion of the investigator will preclude participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Eczema Area and Severity Index (EASI) | at Week 12
  The EASI is a composite score ranging from 0 to 72 that takes into account the degree of erythema, induration/infiltration (papules), excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the percentage of body surface area (BSA) involved for each body region and for the proportion of the body region to the whole body.
  The primary endpoint is the change from baseline in EASI at Week 12.

SECONDARY OUTCOMES:
Change from baseline of Validated Investigator Global Assessment for atopic dermatitis (vIGA-AD) | at Week 12
  The vIGA-AD is a global assessment of the current state of the disease. It is a 5-point morphological assessment of overall disease severity.
Change from baseline of Body Surface Area (BSA) | at Week 12
  The overall BSA affected by disease will be evaluated (from 0% to 100%). The palmar surface of one hand (using the patient's hand and including the fingers) represents 1% of the total BSA.
Change from baseline of Peak pruritus Numerical Rating Scale (NRS) | over 12 weeks
  The intensity of pruritus will be evaluated using a NRS by asking subjects to assign a numerical score representing of the worst intensity over the last 24 hours of their symptoms on a scale from 0 to 10, with 0 indicating no symptoms and 10 indicating the worst imaginable symptoms.
Change from baseline of Facial Eczema Area and Severity Index (EASI) | at Week 12
  The facial EASI is a composite score ranging from 0 to 72 that takes into account the degree of erythema, induration/infiltration (papules), excoriation, and lichenification (each scored from 0 to 3 separately) for each of six facial regions, with adjustment for the percentage of facial surface area involved for each facial region, using the "rule of fours".
Change from baseline of Modified validated Investigator Global Assessment for atopic dermatitis (vIGA-AD) | at Week 12
  The modified vIGA-AD will be used to assess the severity of lesions on the face for subjects with facial erythema at baseline and on the trunk and/or limbs for subjects with atopic dermatitis (AD) on those body parts at baseline.
Change from baseline of the CCL18 Skin Biomarker Level | at Week 12
  The molecular effects of abrocitinib will be evaluated by measuring changes from baseline in CCL18 skin biomarker levels in lesional and nonlesional skin samples.
Change from baseline of the MMP12 Skin Biomarker Level | at Week 12
  The molecular effects of abrocitinib will be evaluated by measuring changes from baseline in MMP12 skin biomarker levels lesional and nonlesional skin samples.
Change from baseline of the Keratin 16 Skin Biomarker Level | at Week 12
  The molecular effects of abrocitinib will be evaluated by measuring changes from baseline in Keratine 16 skin biomarker levels lesional and nonlesional skin samples.
Change from baseline of the S100A7 Skin Biomarker Level | at Week 12
  The molecular effects of abrocitinib will be evaluated by measuring changes from baseline in S100A7 skin biomarker levels lesional and nonlesional skin samples.
Change from baseline of the S100A8 Skin Biomarker Level | at Week 12
  The molecular effects of abrocitinib will be evaluated by measuring changes from baseline in S100A8 skin biomarker levels lesional and nonlesional skin samples.
Change from baseline of the S100A9 Skin Biomarker Level | at Week 12
  The molecular effects of abrocitinib will be evaluated by measuring changes from baseline in S100A9 skin biomarker levels lesional and nonlesional skin samples.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (12):
- United States (6):
  - Inno-6050 Site 22, Birmingham, Alabama
  - Inno-6050 Site 13, Fountain Valley, California
  - Inno-6050 Site 21, Miami Lakes, Florida
  - Inno-6050 Site 19, St. Petersburg, Florida
  - Inno-6050 Site 16, Quincy, Massachusetts
  - Inno-6050 Site 17, Auburn Hills, Michigan
- Canada (6):
  - Inno-6050 Site 15, Winnipeg, Manitoba
  - Inno-6050 Site 18, Newmarket, Ontario
  - Inno-6050 Site 11, Toronto, Ontario
  - Inno-6050 Site 10, Montreal, Quebec
  - Inno-6050 Site 14, Québec, Quebec
  - Inno-6050 Site 20, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No